CLINICAL TRIAL: NCT04685902
Title: Assessing Upper Airway Patency in Tracheostomy Patients During One Way Speaking Valve Trial
Status: Withdrawn | Type: Observational
Why Stopped: Staffing issues
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jie Li, Associate professor, Rush University Medical Center
Other Study IDs: Trach-PMV-001
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Tracheostomy Complication
Keywords: Tracheostomy; Upper airway patency; speaking valve; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with tracheostomy: Adult patients who currently have a tracheostomy and receive an order for one-way speaking valve trial
  Interventions: Device: One-way speaking valve

INTERVENTIONS:
Device: One-way speaking valve — One-way speaking valve is a small device that attaches to the tracheostomy tube, to allows tracheostomy patient to breathe in through his or her trach tube. After the inhalation, the speaking valve closes. Air is breathed out (exhaled) up through the vocal cords, then through the mouth and nose.
  Other Names: Passy muir valve

SUMMARY:
Approximately 24% of ICU patients require the use of a tracheostomy, which impacts vocalization. A one-way speaking valve (SV) can be used to restore vocalization for this patient population. However, if a patient has an obstructed upper airway, SV placement has potential to pose a risk as it might cause asphyxia or even cardiac arrest within minutes, due to the sudden increased intra-thoracic pressure and decreased venous return. Therefore, upper airway patency is crucial in the patient's tolerability and safety to use SV. However, little is available to assess patient's upper airway patency before SV placement. Currently, the predominate way to evaluate readiness is the clinician's subjective assessment based on the quality of vocalization, perceived comfort, and tolerance following SV placement. In the previous in vitro study, the upper airway patency was strongly correlated with the trans-tracheal pressure and the inspiratory flow from upper airway during SV trial. Thus this clinical prospective observational study is aimed to validate the two methods with upper airway patency, which will be validated by bedside ultrasound examination as well.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Current RUMC patient
* An order for a one-way speaking valve trial
* Tracheostomy
* PEEP ≤ 10 cm H2O and FIO2 ≤ 50%
* English speaking

Exclusion Criteria:

* Laryngectomy
* Uncorrected anatomical anomalies
* Unable to communicate
* Hemodynamically unstable
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who currently have a tracheostomy and receive an order for one-way speaking valve trial will be recruited from Rush University Medical Center, Chicago, IL.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Inspiratory flow from upper airway | within 1 minute of measuring patient's inspiratory flow
  Inspiratory flow from upper airway during one-way speaking valve trial
Tidal volume from upper airway | within 1 minute of measuring patient's tidal volume
  Tidal volume from upper airway during one-way speaking valve trial
Tran-tracheal pressure (TTP) | within 15 seconds of measuring TTP
  Tran-tracheal pressure (TTP) during one-way speaking valve trial
leak volume [for mechanically ventilated patients only] | within 1 minute of measuring patient's leak volume
  volume leaked from upper airway during invasive ventilation
Ultrasound results for upper-airway | within 10 minutes of the ultrasound examination
  Ultrasound results include pre-epiglottic space distance/epiglottitis to middle distance of vocal cords (Pre-E/E-VC), thyrohyoid membrane (DSEM), and hyomental distance ratio (HMDR)

SECONDARY OUTCOMES:
Heart rate during one-way speaking valve trial | within 15 minutes of placing one-way speaking valve
  Heart rate during one-way speaking valve trial
Respiratory rate during one-way speaking valve trial | within 15 minutes of placing one-way speaking valve
  Respiratory rate during one-way speaking valve trial
SpO2 during one-way speaking valve trial | within 15 minutes of placing one-way speaking valve
  SpO2 during one-way speaking valve trial
Blood pressure during one-way speaking valve trial | within 15 minutes of placing one-way speaking valve
  Blood pressure during one-way speaking valve trial

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Due to HIPAA, we would not share the individual participant data

REFERENCES:
- [Result] Cheung NH, Napolitano LM. Tracheostomy: epidemiology, indications, timing, technique, and outcomes. Respir Care. 2014 Jun;59(6):895-915; discussion 916-9. doi: 10.4187/respcare.02971. PMID 24891198
- [Result] Johnson DC, Campbell SL, Rabkin JD. Tracheostomy tube manometry: evaluation of speaking valves, capping and need for downsizing. Clin Respir J. 2009 Jan;3(1):8-14. doi: 10.1111/j.1752-699X.2008.00100.x. PMID 20298366
- [Result] Singh RK, Saran S, Baronia AK. The practice of tracheostomy decannulation-a systematic review. J Intensive Care. 2017 Jun 20;5:38. doi: 10.1186/s40560-017-0234-z. eCollection 2017. PMID 28649385
- [Result] Falcetta S, Cavallo S, Gabbanelli V, Pelaia P, Sorbello M, Zdravkovic I, Donati A. Evaluation of two neck ultrasound measurements as predictors of difficult direct laryngoscopy: A prospective observational study. Eur J Anaesthesiol. 2018 Aug;35(8):605-612. doi: 10.1097/EJA.0000000000000832. PMID 29889671